CLINICAL TRIAL: NCT04117061
Title: Optimizing the Diagnosis of Acute Appendicitis - Open, Randomized, Parallel Groups, Prospective Clinical Trial
Brief Title: Optimizing the Diagnosis of Acute Appendicitis
Acronym: OPTIMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Tomas Poskus, Profesor at Vilnius University, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UADO-1
Record Dates: First submitted 2019-06-29; First posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Observation

STUDY DESIGN:
Intervention Model Description: Open, randomized, parallel groups prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patient gets usual diagnostic path: after inconclusive ultrasound is refered to CT scan.
- Observation (Active Comparator): Patient after inconclusive primary evaluation is observed in emergency room for 8-12 hours and after the clinical evaluation, laboratory results and ultrasound examination is repeated.
  Interventions: Procedure: Observation

INTERVENTIONS:
Procedure: Observation — Patient after primary investigation is observed for 8-12 hours, (instead of being send directly to CT scan), after observation repeated clinical evaluation, laboratory tests and ultrasound examination are done , if final diagnosis stays unclear the patient is refered to CT scan.
  Arms: Observation

SUMMARY:
Aim of the study: to identify the signs of acute appendicitis delta signs - clinical, laboratory or ultrasound signs, whose change (delta) would allow to identify or deny the diagnosis of acute appendicitis without a computed tomography examination and thus to lower computed tomography rates.

DETAILED DESCRIPTION:
This study consists of two parts:

* In the first part investigators enroll all patients (except pregnant) that are refered to Vilnius University Hospital Santaros clinics with suspected acute appendicitis in order to get cohort data. All patient get primary clinical evaluation, laboratory tests (WBC, CRP) an ultrasound examination.
* After primary evaluation if final diagnosis could not be made, and investigator still suspect acute appendicitis, participant is included in to randomised study part.
* Randomised sudy part has two arms: control and observation groups.
* Control group get the traditional diagnostic path - is refered to CT scan examination.
* Observation group get repeated evaluation after 8-12 hours and only than is diagnosis stays unclear, patient gets a CT scan.
* All patient are contacted after 30 days after visit to our hospital, to get information about their health status and possible additional visits to other hospitals or operations.

ELIGIBILITY:
Inclusion Criteria:

* Patient with the symptoms of acute appendicitis: pain in the right lower quadrant, pain migration from epigastrium to right lower quadrant, nausea, rebound pain, elevated temperature.

Exclusion Criteria for randomized part:

* Pregnant patient.

Inclusion Criteria for randomized part:

* After primary clinical, laboratory and ultrasound examination diagnosis of acute appendicitis could not be confirmed or excluded.
* No other gynecological, urological ir gastroenterological pathology is confirmed.

Exclusion Criteria for randomized part:

* Clinical symptoms lasts for longer than 48 hours
* Signs of peritonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of the CT scans number | 24 hours
  when performing alternative diagnostic protocol, that includes patient observation for short period we expect to reduce a number of CT scans performed, for the patients with suspected acute appendicitis.
Negative appendectomy rate | 30 days
  We expect the negative appendectomy rate will will not increase while using alternative diagnostic protocol that includes patient observation.

SECONDARY OUTCOMES:
Delta marker White blood cell count | 12 hours
  The changes in white blood cell count over the time that might show higher or lower probability of possible acute appendicitis.
Delta marker CRP count | 12 hours
  The changes CRP level over the time that might show higher or lower probability of possible acute appendicitis.
Delta marker Alvarado acute appendicitis risk evaluation score | 12 hours
  Delta marker Alvarado acute appendicitis risk evaluation score Tha changes in score over the time that might show higher or lower probability of possible acute appendicitis. Scale ranges decribe a prediction of having acute appendicitis: 1-4 33 % of having appendicitis, 5-6 66 % of hanving, 7-10 93 % of having appendicitis.
Delta marker changes in ultrasound results | 12 hours
  The changes in ultrasound findings over the time may progress and influence investigator to change opinion about the concusion. Repeated ultrasound diagnosis might change from unequivocal to acute apendicitis (and CT scan can be avoided then). We do use structured conclusions of the ultrasound exam, that might be: accute appendicitis; apendix visualised but changes are equivocal; apendix visualised uninflamed; apendix not visualised, but there are secondary findings; apendix not visualised and there is no secondary findings. We are going to measure the change in final ultrasound diagnosis over the time.
'Appendicitis Inflammatory Response (AIR) Score' | 12 hours
  'Appendicitis Inflammatory Response (AIR) Score') evaluates the risk for acute appendicitis. scale ranges are: 0-4 low probability outpatient follow up, 5-8 inermediate probability in hospital observation, 9-12 high probability, surgical treatment..

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Poskus, Professor, Principal Investigator — Vilnius University, Faculty of medicine, Institute of clinical medicine
Locations (1):
- Faculty of medicine, Institue of clinical medicine, Clinic of gastroenterology, nephrourology and surgery, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No
There are no future intensions make IPD available.